CLINICAL TRIAL: NCT04535661
Title: A Retrospective Single Center Study of the Risk Factors for Colonization or Infection With Carbapenem-Resistant Enterobacteriaceae in PICU Hospitalized Children
Brief Title: Risk Factors for Colonization or Infection With Carbapenem-Resistant Enterobacteriaceae in Children
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-05
Record Dates: First submitted 2020-08-26; First posted 2020-09-02 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non CRE: Children with a negative culture for CRE during their stay in PICU are defined as non CRE.
- CRE colonization: Children who have a positive culture for CRE during their stay in PICU but lack of clinical symptoms are defined as CRE colonization.
- CRE infection: Children who have a positive culture for CRE during their stay in PICU combined with clinical symptoms are defined as CRE infection.

SUMMARY:
Carbapenem-resistant Enterobacteriaceae (CRE) are increasingly identified in children in China. Pediatric intensive care unit (PICU) is the high-risk area. However, data on the epidemiology of CRE in hospitalized children in PICU are limited. The objectives of this study are to characterize the risk factors for colonization or infection with CRE and describe the microbiologic characteristics of pediatric CRE isolates. The investigators will perform a single retrospective study from January 2018 to December 2019 at PICU of Children's Hospital of Fudan University .

DETAILED DESCRIPTION:
The investigators intend to enroll all children who were hospitalized in pediatric intensive care unit PICU of Children's Hospital of Fudan University from January 2018 to December 2019. Children who had positive cultures for any Enterobacteriaceae species before their admission will be excluded. Children with a PICU length of day less than 48h will also be excluded. According to their clinical cultures results, they will be divided into non-CRE、CRE colonization and CRE infection. CRE was defined according to the 2015 Centers for Disease Control and Prevention (CDC) definition as an isolate resistant to imipenem, meropenem, or ertapenem. Clinical and demographic data will be collected from the electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* All children hospitalized in PICU of Children's Hospital of Fudan University from January 2018 to December 2019.

Exclusion Criteria:

* discharge within 48 hours
* patients had a positive culture for CRE before admission
* incomplete clinical and demographic data

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children hospitalized in PICU of Children's Hospital of Fudan University from January 2018 to December 2019
Sampling Method: Non-Probability Sample
Enrollment: 536 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality | within 28 days after they discharged from PICU
  The death rate of children in 28 days after their discharged from PICU

SECONDARY OUTCOMES:
length of stay in PICU | within 28 days after they discharged from PICU
  Time from PICU admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gangfeng Yan, Principal Investigator — Children's Hospital of Fundan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided